CLINICAL TRIAL: NCT04929405
Title: Pilot-Testing a Theoretically Based Digital Intervention for Bereaved Parents (ADAPT)
Brief Title: Pilot Testing ADAPT a Bereavement Care Intervention
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Palliative Care Research Cooperative Group (Network); Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Nancy Dias, Assistant Professor, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCIRB 19-001984
Record Dates: First submitted 2020-08-25; First posted 2021-06-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Bereavement
Keywords: Bereavement; Palliative Care; Web-based Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): This group has access to the intervention (website for bereaved parents)
  Interventions: Behavioral: ADAPT

INTERVENTIONS:
Behavioral: ADAPT — ADAPT, is multi-modal to promote a targeted approach to individual parental bereavement experiences and is not time or geographically limited. ADAPT is based on the theoretical foundations of the Adaptive Leadership (AL) framework. Our interdisciplinary team developed a web-based, multi-modal intervention, labeled ADAPT, that incorporates varied self-management strategies including: A: Asking for assistance (option to connect with child's healthcare team); DA: Developing Adaptive ability (self-management tools: e.g. stress reduction, legacy building); P: Accessing Pertinent online resources (grief support networks/websites); and T: Tracking one's health (self-administered surveys for grief, sleep, anxiety, and depression). Parents can download ADAPT on any digital device (phones/computers) using a Quick Response (QR) bar code or weblink.

SUMMARY:
Parental bereavement experiences are unique and require interventions adaptable to individual experiences.The web-based, multi-modal intervention, labeled ADAPT, incorporates varied self-management strategies including: A: Asking for assistance (option to connect with child's healthcare team); DA: Developing Adaptive ability (self-management tools: e.g. stress reduction, legacy building); P: Accessing Pertinent online resources (grief support networks/websites); and T: Tracking one's health (self-administered surveys for grief, sleep, anxiety, and depression). A quasi-experimental, treatment-only design will be used for this study. The hypothesis is that the ADAPT intervention will promote positive adaptation to influence grief integration and consequently affect health outcomes (improved sleep and social interactions, and decreased anxiety and depressive symptoms).The purpose of this study is to describe the nature and degree of clinical benefit of the intervention on bereaved parents' health outcomes.

DETAILED DESCRIPTION:
ADAPT, is multi-modal intervention that promotes a targeted approach to individual parental bereavement experiences. ADAPT is based on the theoretical foundations of the Adaptive Leadership (AL) framework. ADAPT, incorporates varied self-management strategies including: A: Asking for assistance (option to connect with child's healthcare team); DA: Developing Adaptive ability (self-management tools: e.g. stress reduction, legacy building); P: Accessing Pertinent online resources (grief support networks/websites); and T: Tracking one's health (self-administered surveys for grief, sleep, anxiety, and depression). Parents can download ADAPT on any digital device (phones/computers) using weblink.

B. Study Purpose and Objective(s)

The purpose of this study is to describe the nature and degree of clinical benefit of the intervention on bereaved parents' health outcomes. The Specific Aims are:

Aim 1: Assess the acceptability and feasibility of the ADAPT intervention components. Acceptability will be assessed with a modified standardized acceptability survey and cognitive interviews. Feasibility will be assessed by accrual (recruitment), attrition, and intervention engagement (i.e., frequency, duration, and interaction). Intervention engagement data will be obtained via Google analytics and cognitive interviews.

Hypothesis 1.1: ADAPT is acceptable to participants (> 80% acceptability based on survey).

Hypothesis 1.2: Delivery of ADAPT is feasible in terms of accrual (N=30), attrition (15%), and intervention engagement (minimally accessed 3 times for >15 minutes and used at least 2 self-management strategies) Aim 2: Determine if the use of the ADAPT intervention components results in a clinically meaningful change in grief integration (Brief Grief Questionnaire) and bereaved parents' health outcomes (Visual Analogue Scale for overall health and PROMIS surveys for sleep, social isolation, anxiety, and depression). Hypothesis 2.1: After completing the ADAPT intervention, participants will demonstrate improvement in health outcome scores when compared to baseline (T0).

Design: quasi-experimental, treatment-only design. Sample: N=35 parents of children who have died while being followed for care at either Akron Children's Hospital or Cardinal Glennon Children's hospital.

Recruitment: Participants will be recruited into two groups. Group 1 will be parents whose child died 4 weeks (+ 2 weeks) prior; Group 2 will be parents whose child died three months (+/- 2 weeks) prior to enrollment. Either a mother or a father for any one child will be recruited.

For both the groups, a Study Information Sheet will be included in each bereavement packet sent or mailed home, at either 4 week (group 1) or 3 months (group 2) after the child has died. This Study Information Sheet will have a study-specific phone number and email address for a clinical research coordinator, through which the parent can immediately opt in or opt out. If there is no response following one to two weeks after the bereavement packet was sent, the bereaved parents will be contacted by study staff via telephone to assess interest, discuss the study, and answer any questions they may have. If the parent agrees to participate, econsent will be completed using REDCap. After completing the econsent, participants will have access to ADAPT and will be provided a REDCap survey link to allow self-completion of baseline questionnaires (T0) (see Table 1). Three months after completing the intervention (T1), participants will again be provided a REDCap survey link to post-intervention questionnaires (see Table.1). At that time, a semi-structured cognitive interview with participants will be scheduled. The interviews will be conducted via telephone and will be recorded, transcribed, and verified for accuracy by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent and legal guardian of a deceased child who was 18 years old or younger at time of death
* Cause of death of the deceased child is illness
* Parent age 18 years or older at time of child's death
* Ability to speak and read English sufficient to participate in the study

Exclusion Criteria:

* Step-, foster-, grand- or fictive parent of a child who has died
* Deceased child was unborn or over age 18 years at time of death
* Deceased child was in legal custody of county or state jurisdiction
* Cause of child's death was in utero or traumatic
* Parent age less than 18 years
* Inability to speak and read English sufficient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | 3 months
  Recruited 35 participants in the study timeframe
Retention | 3 months
  Participants complete surveys at pre and post intervention.

SECONDARY OUTCOMES:
Sleep | 3 months
  Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) sleep scores from baseline to 3 months. The final score for these PROMIS measures is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scoring will be completed by uploading deidentified data to the Health Measures Scoring Service using the General and Clinical reference population.
Grief | 3 months
  Change in grief scores of the Brief Grief Questionnaire from baseline to 3 months. If the participants score 4 or above they need full evaluation.
Social isolation | 3 months
  Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) social isolation scores from baseline to 3 months. The final score for these PROMIS measures is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scoring will be completed by uploading deidentified data to the Health Measures Scoring Service using the General and Clinical reference population.
Anxiety | 3 months
  Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scores from baseline to 3 months. The final score for these PROMIS measures is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scoring will be completed by uploading deidentified data to the Health Measures Scoring Service using the General and Clinical reference population.
Depression | 3 months
  Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) depression scores from baseline to 3 months. The final score for these PROMIS measures is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scoring will be completed by uploading deidentified data to the Health Measures Scoring Service using the General and Clinical reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Dias, PhD, Principal Investigator — East Carolina University
Locations (2):
- United States (2):
  - Cardinal Glennon Childrens Hospital, St Louis, Missouri
  - Akron Children's Hospital, Akron, Ohio

IPD SHARING:
Plan to Share IPD: No